CLINICAL TRIAL: NCT01571492
Title: Continuous L2 Paravertebral Block Versus Continuous Lumbar Plexus Block for Postoperative Analgesia After Total Hip Arthroplasty
Brief Title: Continuous L2 Paravertebral Block Versus Continuous Lumbar Plexus Block for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jacques E. Chelly, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO09010511
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Total Hip Arthroplasty
Keywords: Postoperative Pain; Nerve block; Total Hip Arthroplasty; Postoperative analgesia; Lumbar Plexus Catheters; L2 Paravertebral Catheters
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L2 Paravertebral peripheral nerve block (Experimental): L2 paravertebral peripheral nerve block catheter will be placed.
  Interventions: Procedure: L2 Paravertebral catheter nerve block
- Continuous Lumbar plexus peripheral nerve block (Active Comparator): Continuous unilateral lumbar plexus peripheral nerve block catheter will be placed.
  Interventions: Procedure: Continuous Lumbar plexus nerve block

INTERVENTIONS:
Procedure: L2 Paravertebral catheter nerve block — A continuous L2 paravertebral catheter will be placed according to UPMC standard of care practices.
  Arms: L2 Paravertebral peripheral nerve block
Procedure: Continuous Lumbar plexus nerve block — A continuous unilateral lumbar plexus catheter will be placed according to UPMC standard of care practices.
  Arms: Continuous Lumbar plexus peripheral nerve block

SUMMARY:
This prospective study is intended to compare the analgesic efficacy, preservation of lower extremity motor power and side-effect profile of L2 Paravertebral lumbar plexus approach compared to Posterior nerve stimulation guided lumbar plexus approach, continuous local anesthetic infusion postoperative analgesia of Total Hip Arthroplasty.

The L2 Paravertebral technique of lumbar plexus block, as part of a multimodal pain treatment, could be a cost-effective alternative with a equal profile of analgesic efficacy and motor power sparing with greater promotion of early achievement of postoperative physical therapy goals.

DETAILED DESCRIPTION:
The nerve stimulator guided technique of continuous lumbar plexus block (LPB) is the accepted standard of care at University of Pittsburgh Medical Center (UPMC) for the management of postoperative analgesia after Total Hip Arthroplasty. Over 900 continuous lumbar plexus blocks were performed at UPMC Presbyterian Shadyside hospital within the last year alone. Continuous thoracic paravertebral block (TPVB) is also commonly performed at UPMC Presbyterian Shadyside . Over 2000 are performed annually for a wide variety of surgical procedures. Recently authors have suggested that a lumbar paravertebral block (LPVB) may represent an alternative approach to the lumbar plexus. Indeed the L2 paravertebral approach of the lumbar plexus has been described to provide adequate postoperative analgesia following hip arthroscopic surgery. However, to date, there is no prospective direct comparison between L2 Lumbar plexus approach and the posterior approach for postoperative analgesia after Total Hip Arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* No contraindications to placement of a lumbar plexus posterior block or paravertebral block.
* ASA status I-III
* Scheduled for open total hip arthroplasty with the same surgeon.
* Patients without painful conditions or chronic use of opioid or antineuropathic medications.
* Patient who are not expected to receive therapeutic anticoagulation in the postoperative period.
* No Known allergies to the medications used in the study.
* Patients willing to receive spinal anesthesia

Exclusion Criteria:

* Age under 18 years or older than 75 years.
* Any contraindication to a placement of continuous lumbar plexus Block.
* American Society of Anesthesiologist physical status IV or greater.
* Chronic painful conditions.
* Preoperative opioid tolerant use.
* Coagulation Abnormalities or patients who are expected to be on therapeutic anticoagulants postoperatively.
* Allergy to any of the drugs/agents used study protocol.
* Personal or family history of malignant hyperthermia.
* Serum creatinine greater than 1.4 mg/dl.
* Pregnancy
* Having an altered mental status (not oriented to place, person, or time)
* Any comorbid condition that, in the judgment of the consulting orthopedic surgeon, or intraoperative anesthesiologist, would proscribe the patient from any aspect of the study.
* Patient refusal.
* Lumbar plexus block performed with loss of resistance technique
* Patient requiring postoperative management in the ICU

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Opiate consumption | 24 postoperatively
  Postoperative Opiate consumption will be recorded as Morphine IV mg equivalent, for the first 24 hours.

SECONDARY OUTCOMES:
NRS Pain Score (at rest) | 24 and 48 hours postoperatively
  Pain scores at Rest will be recorded at 24 and 48 Hours
NRS Pain Score during physical therapy | 24 and 48 hours postoperatively
  Pain scores at Rest and During physical therapy will be recorded at 24 and 48 Hours
TUG (Timed Up and Go) | 24 hours postoperatively
  The timed get up and go test is a measurement of mobility. It includes a number of tasks such as standing from a seating position, walking, turning, stopping, and sitting down which are all important tasks needed for a person to be independently mobile.
Straight Leg Raise(SLR) | 24 hours postoperatively
  In supine position with the extremity being tested and contralateral flexed LE with foot flat on surface. Patient is instructed to lift extremity to level of contralateral knee. Inability to lift entire LE off of the surface to the level of the contralateral knee would be indicative of hip flexor weakness. If the patient is able to lift LE off of the surface, however the knee flexes/unable to maintain full knee extension, this is indicative of quad weakness.
Long arc quad (LAQ) | 24 hours postoperatively
  In sitting position at the edge of the bed or chair. Patient is asked to extend lower leg fully on side that is being tested. If able, this is indicative that quad function is intact. If unable to fully extend knee, would indicate quad weakness.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Marino J, Russo J, Kenny M, Herenstein R, Livote E, Chelly JE. Continuous lumbar plexus block for postoperative pain control after total hip arthroplasty. A randomized controlled trial. J Bone Joint Surg Am. 2009 Jan;91(1):29-37. doi: 10.2106/JBJS.H.00079. PMID 19122076
- [Background] Lee EM, Murphy KP, Ben-David B. Postoperative analgesia for hip arthroscopy: combined L1 and L2 paravertebral blocks. J Clin Anesth. 2008 Sep;20(6):462-5. doi: 10.1016/j.jclinane.2008.04.012. PMID 18929290
- [Background] Capdevila X, Macaire P, Dadure C, Choquet O, Biboulet P, Ryckwaert Y, D'Athis F. Continuous psoas compartment block for postoperative analgesia after total hip arthroplasty: new landmarks, technical guidelines, and clinical evaluation. Anesth Analg. 2002 Jun;94(6):1606-13, table of contents. doi: 10.1097/00000539-200206000-00045. PMID 12032037
- [Background] Siddiqui ZI, Cepeda MS, Denman W, Schumann R, Carr DB. Continuous lumbar plexus block provides improved analgesia with fewer side effects compared with systemic opioids after hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):393-8. doi: 10.1016/j.rapm.2007.04.008. PMID 17961837
- [Background] Chudinov A, Berkenstadt H, Salai M, Cahana A, Perel A. Continuous psoas compartment block for anesthesia and perioperative analgesia in patients with hip fractures. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):563-8. doi: 10.1016/s1098-7339(99)90050-0. PMID 10588563
- [Background] Kaloul I, Guay J, Cote C, Fallaha M. The posterior lumbar plexus (psoas compartment) block and the three-in-one femoral nerve block provide similar postoperative analgesia after total knee replacement. Can J Anaesth. 2004 Jan;51(1):45-51. doi: 10.1007/BF03018546. PMID 14709460
- [Background] Farny J, Drolet P, Girard M. Anatomy of the posterior approach to the lumbar plexus block. Can J Anaesth. 1994 Jun;41(6):480-5. doi: 10.1007/BF03011541. PMID 8069987
- [Background] Ilfeld BM, Ball ST, Gearen PF, Le LT, Mariano ER, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Meyer RS. Ambulatory continuous posterior lumbar plexus nerve blocks after hip arthroplasty: a dual-center, randomized, triple-masked, placebo-controlled trial. Anesthesiology. 2008 Sep;109(3):491-501. doi: 10.1097/ALN.0b013e318182a4a3. PMID 18719448
- [Background] Mannion S, O'Callaghan S, Walsh M, Murphy DB, Shorten GD. In with the new, out with the old? Comparison of two approaches for psoas compartment block. Anesth Analg. 2005 Jul;101(1):259-64, table of contents. doi: 10.1213/01.ANE.0000153866.38440.43. PMID 15976242
- [Background] Williams BA, Murinson BB. Diabetes mellitus and subclinical neuropathy: a call for new paths in peripheral nerve block research. Anesthesiology. 2008 Sep;109(3):361-2. doi: 10.1097/ALN.0b013e3181829f0d. No abstract available. PMID 18719433
- [Background] Zink W, Sinner B, Zausig Y, Graf BM. [Myotoxicity of local anaesthetics: experimental myth or clinical truth?]. Anaesthesist. 2007 Feb;56(2):118-27. doi: 10.1007/s00101-006-1121-5. German. PMID 17235544